CLINICAL TRIAL: NCT07404618
Title: Development and Preliminary Testing of a Peer Narrative Video Intervention for Older Adults With Chronic Pain
Brief Title: Video Intervention for Older Adults With Chronic Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2408-001; RF1AG089083 (NIH)
Record Dates: First submitted 2026-02-05; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Chronic Pain; Musculoskeletal Pain; Older Adults With Chronic Pain
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reclaim Your Day (Experimental): Reclaim You Day is a 6-part video intervention that features peers with lived experience describing how they learned to live well with their chronic pain and is provided for 6 weeks.
  Interventions: Behavioral: Reclaim Your Day
- Health education (Active Comparator): Health education is a 6-part video series covering various health topics and is offered over 6 weeks.
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: Reclaim Your Day — Reclaim You Day is a 6-part video intervention that features peers with lived experience describing how they learned to live well with their chronic pain and is provided for 6 weeks.
  Arms: Reclaim Your Day
Behavioral: Health education — Health education is a 6-part video series covering various health topics and is offered over 6 weeks.
  Arms: Health education

SUMMARY:
Chronic musculoskeletal (MSK) pain, which includes spinal pain, osteoarthritis, and fibromyalgia, is a common and costly problem for older adults and is associated with decreased quality of life. In this project, we propose to create Reclaim Your Day (RYD), which will consist of 6, 30-min weekly video episodes highlighting patients' inspiring and illustrative experiences living with chronic pain in order to teach current patients with chronic MSK pain how to apply ACT's evidence-based strategies. We will conduct a pilot RCT (n=100) of older adults with chronic MSK pain. All participants will receive an introductory pain education video. Participants will be randomized to receive either RYD or a comparison intervention (health education videos). We will examine RYD feasibility and acceptability as well as changes over time in outcomes (pain interference, depression, quality of life) and putative mediators.

DETAILED DESCRIPTION:
Chronic musculoskeletal (MSK) pain, which includes spinal pain, osteoarthritis, and fibromyalgia, is a common and costly problem for older adults and is associated with decreased quality of life. There is a clear need for interventions that increase one's ability to cope with chronic pain and engage in meaningful life activities even with the presence of chronic pain. Acceptance and Commitment Therapy (ACT) is a psychotherapy that uses mindfulness and psychological acceptance to support individuals in working toward behavioral goals guided by their personal values, even in the presence of undesirable experiences such as chronic pain. Clinical practice guidelines recommend the use of ACT for treating chronic pain based on evidence of effectiveness from multiple RCTs. However, uptake and reach are limited because there are insufficient numbers of mental health professionals who currently offer ACT or other recommended therapies (e.g., cognitive-behavioral therapy) for chronic pain. In addition, many older adults are not willing or able to engage in traditional psychotherapy for chronic pain even when it is available. Although some bibliotherapy and digital health interventions (e.g., apps) have been developed for treating pain, many older adults fail to use them due to low levels of comfort with technology or lack of motivation for intensive self-guided approaches. Narrative communication is an alternative way to deliver behavior change principles that involves "storytelling" involving real patients talking about their struggles and recovery progress. Therapeutic narratives delivered via videos may be more engaging and immersive than traditional self-help formats for older adults. In this project, we propose to create Reclaim Your Day (RYD), which will consist of 6, 30-min weekly video episodes highlighting patients' inspiring and illustrative experiences living with chronic pain in order to teach current patients with chronic MSK pain how to apply ACT's evidence-based strategies. We will conduct a pilot RCT (n=100) of older adults with chronic MSK pain. All participants will receive an introductory pain education video. Participants will be randomized to receive either RYD or a comparison intervention (health education videos). We will examine RYD feasibility and acceptability as well as changes over time in outcomes (pain interference, depression, quality of life) and putative mediators.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic MSK pain. Consistent with existing guidance, the experience of pain must be present most days of the week over the past 3 months, of at least moderate intensity.
2. Pain interferes with everyday activities.
3. Age 55 or older.
4. Proficiency in English sufficient to engage in informed consent and understand assessments and materials.
5. Reliable internet access.

Exclusion Criteria:

1. Currently receiving acceptance/mindfulness or similar psychotherapy for chronic pain management.
2. Current severe substance use problems.
3. Cognitive impairment that would interfere with a person's capacity to complete the study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire (CSQ) | 6 weeks
  The Client Satisfaction Questionnaire (CSQ) is an 8 item self-report measure of patient satisfaction with treatment. The total score will be used and ranges from 8 to 32 with higher scores indicating greater satisfaction with treatment.

SECONDARY OUTCOMES:
Brief Pain Inventory (BPI) - Pain Interference subscale | 6 weeks
  The Brief Pain Inventory (BPI) - Pain Interference subscale is a 7-item patient-reported rating of how much pain interferes with daily functioning on 0-10 numeric scales and is typically scored as the mean of the 7 items (range 0-10, higher scores = greater interference).

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Gaudiano, PhD, Principal Investigator — Butler Hospital; Lisa Uebelacker, PhD, Principal Investigator — Butler Hospital

IPD SHARING:
Plan to Share IPD: Yes
We will deposit data in the National Archive of Computerized Data on Aging (NACDA), which is supported by NIA and is part of the Inter-university Consortium for Political and Social Research (ICPSR).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be archived by the anticipated end of the study date.
Access Criteria: These files, in which direct and indirect identifiers have been removed to minimize disclosure risk, may be accessed directly through the ICPSR website. After agreeing to Terms of Use, users with an ICPSR MyData account and an authorized IP address from a member institution may download the data, and non-members may purchase the files.
URL: https://www.icpsr.umich.edu/sites/icpsr/home